CLINICAL TRIAL: NCT06094023
Title: Development and Validation of Food Frequency Questionnaire to Assess the Dietary Intake of Folic Acid and Vitamin B12 Among Teenage Girls in South Ethiopia.
Brief Title: Dietary Intake of Folic Acid and Vitamin B12 Among Teenage Girls - Validation of Food Frequency Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Arba Minch University (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Addis Ababa University (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0137-A
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dietary Assessment
Keywords: Dietary assessment; Food Frequency Questionnaire; Multi-pass 24 hour food recall; Semi-quantitative; Vitamin B12; Folic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teenage girls between 13 and 19 years living in the Arba Minch Demographic and Surveillance site.: Participants in this study should be acquainted with cooking practices to be able to cite all the ingredients that are used in the preparation of the dishes/ meals
  Interventions: Other: Food Frequency Questionnaire; Other: 24 Hour food recall

INTERVENTIONS:
Other: Food Frequency Questionnaire — Food frequency questionnaires (FFQs) are a common method for measuring dietary intake in large epidemiological studies, in particular in low literacy settings were diaries and food history would not be viable.
Other: 24 Hour food recall — Standardized and validated approach of collecting all foods, beverages, and supplements consumed during the past 24 hours.

SUMMARY:
Folate and vitamin B12 deficiencies are associated with various health issues, including anemia, cardiovascular disease, depression, and birth defects. Accurate and objective estimates of dietary intake are necessary to assess any effects of nutritional status in epidemiologic studies. This study aims to develop and validate a three-month semi-quantitative food frequency questionnaire for the assessment of dietary intake of folic acid and vitamin B12, against four*two multiple-pass 24-hr dietary recall among teenage girls in South Ethiopia

DETAILED DESCRIPTION:
Folic acid and vitamin B12 play an interdependent role in key cellular processes, namely deoxyribonucleic acid synthesis, cell division, red blood cell formation, and nervous system myelination. Folic acid is an essential nutrient in the growth and development of the cerebral cortex. It promotes the thickness of the cerebral cortex; which is directly proportional to the intelligence quotient, the neurocognitive and psychological development of the child. Both folate and vitamin B12 participate in the conversion of homocysteine to methionine, such that a deficiency in either vitamin will result in elevated serum concentrations of homocysteine where high levels of serum homocysteine are associated with an increased risk for depression. Deficiencies in folate and vitamin B12 have been shown to delay growth spurt and pubertal growth during adolescence. Some studies also showed that there is an association between overweight and obesity with lower serum vitamin B12 and folate levels.

In research, there are several challenges in the accurate assessment of diet and nutrition. In the Ethiopian context, there is no tool that specifically assesses dietary intake of folic acid and vitamin B12 in adolescents. In this project, reliable dietary assessment tools for assessing dietary intake of folic acid and vitamin B12 will be developed and validated for future use as an unbiased reference measure. The dietary validation study will start by conducting a food frequency questionnaire (FFQ). The FFQ will consider the recall time frame of the previous three months assuming that the consumption patterns for folate and vitamin B12-rich foods of participants over a three-month period can be considered as their usual food intake. The FFQ will be administered to the selected study participants four times: at the beginning of the validation study, after 3 and 6 months, and at 9 months (the end of the study). The same participants will be also asked to complete two 24-hour food recalls every three months in a nine-month period. The first 24-hour recall questionnaires will be collected at least one week after the first FFQ, and one within the 3-month period considering one weekday and one weekend day. A total of eight 24-hour food recalls and four FFQs will be collected.

Study objective

The objective of this sub study is to develop and validate a FFQ that can be used to assess the dietary intake of folic acid and vitamin B12 among teenage girls who reside in rural communities of Arba Minch Health and Demographic Surveillance Sites (AM-HDSS), South Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* One or both of their parents signed an informed consent form and the girls agreed.
* Their parents and the girl planned to stay during the period of the study (minimum 9 months) in the kebele.
* Aged between 13 and 19 years
* Familiar with the diet and cooking practices
* Accept enumerators for home visit and data collection for one year

Exclusion Criteria:

* Teenage girls who are pregnant and/or are lactating

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted among randomly selected teenage girls between the age of 13-19 years who resides in households at AM-HDSS. The data collection will be done at the selected teenagers' households.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
1. Mean/Median proportion of folic acid intake assessed by the 24 hour recalls | 12 month
  Mean/Median proportion of folic acid intake from (Cereal and cereal products, Tubers & Roots, Legumes & Legume products, Vegetables, Fruit & Berries, Meat & Poultry, Fish, Dairy products, Egg, Sugars, Oil, Fat, Oil seeds & nuts, Herbs & spices , soft drinks and beverages) assessed by 24 hour recalls The recommended intake for folic acid for teenage girls aged between 13 and 19 years is set at 400 micrograms/day
2. Mean/median proportion of folic acid intake assessed by the food frequency questionnaire | 12 month
  Mean/Median proportion of folic acid intake from (Cereal and cereal products, Tubers & Roots, Legumes & Legume products, Vegetables, Fruit & Berries, Meat & Poultry, Fish, Dairy products, Egg, Sugars, Oil, Fat, Oil seeds & nuts, Herbs & spices , soft drinks and beverages) assessed by food frequency questionnaire.
  The recommended intake for folic acid for teenage girls aged between 13 and 19 years is set at 400 micrograms/day
3. Mean/median proportion of vitamin B12 intake assessed by the 24 hour recalls | 12 month
  Mean/Median proportion of vitamin B12 intake from (Meat & Poultry, Fish, Dairy products, Egg, soft drinks and beverages) assessed by 24 hour recalls
  The recommended intake for vitamin B12 for teenage girls aged between 13 and 19 years is set at 2.4 micrograms/day
4. Mean/median proportion of vitamin B12 intake assessed by the food frequency questionnaire | 12 month
  Mean/Median proportion of vitamin B12 intake from (Meat & Poultry, Fish, Dairy products, Egg, soft drinks and beverages) assessed by food frequency questionnaire
  The recommended intake for vitamin B12 for teenage girls aged between 13 and 19 years is set at 2.4 micrograms/day

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, MD. PhD, Principal Investigator — University Ghent
Locations (1):
- Arba Minch University, Arba Minch, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes and its Panel on Folate, Other B Vitamins, and Choline. Dietary Reference Intakes for Thiamin, Riboflavin, Niacin, Vitamin B6, Folate, Vitamin B12, Pantothenic Acid, Biotin, and Choline. Washington (DC): National Academies Press (US); 1998. Available from http://www.ncbi.nlm.nih.gov/books/NBK114310/ PMID 23193625
- [Background] Beydoun MA, Shroff MR, Beydoun HA, Zonderman AB. Serum folate, vitamin B-12, and homocysteine and their association with depressive symptoms among U.S. adults. Psychosom Med. 2010 Nov;72(9):862-73. doi: 10.1097/PSY.0b013e3181f61863. Epub 2010 Sep 14. PMID 20841559